CLINICAL TRIAL: NCT03825744
Title: A Phase III Multicenter Randomized Study of Hetrombopag or Placebo in Treatment-Naive Severe Aplastic Anemia
Brief Title: Hetrombopag or Placebo in Treatment-Naive Severe Aplastic Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-TPO-SAA-III
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-01

CONDITIONS: Severe Aplastic Anemia
Keywords: SAA
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hetrombopag Olamine+Standard Therapy (Experimental)
  Interventions: Drug: Hetrombopag Olamine+Standard Therapy
- Placebo+Standard Therapy (Placebo Comparator)
  Interventions: Drug: Placebo+Standard Therapy

INTERVENTIONS:
Drug: Hetrombopag Olamine+Standard Therapy — once daily
  Arms: Hetrombopag Olamine+Standard Therapy
Drug: Placebo+Standard Therapy — once daily
  Arms: Placebo+Standard Therapy

SUMMARY:
This is a multicenter, randomized, placebo-control, phase III study to investigate hetrombopag in subjects with severe AA who are treated naive.

180 treated naive patients with SAA will be enrolled in the study. The primary objective of the study will be the rate of complete hematologic response at six months.

ELIGIBILITY:
Inclusion Criteria:

1.15 Years to 75 Years (weight greater than 50 kg if Age < 18 years old). 2.Severe aplastic anemia characterized by Bone marrow cell proliferation less than 25 percent (If ≥25% but <50%, the remaining hematopoietic cells should be <30%) AND At least two of the following: Absolute neutrophil count <0.5×109/L; Platelet count <20×109/L; Absolute reticulocyte count <20×109/L.

3.Unsuitable or unwilling to perform hematopoietic stem cell transplantation (HSCT).

4.Signed informed consent.

Exclusion Criteria:

1. Diagnosis of whole blood cell reduction due to other causes or bone marrow hypoproliferative diseases.
2. Subjects who have previously received immunosuppressive therapy with mycophenolate mofetil, sirolimus, high dose cyclophosphamide (≥45mg/kg/d), alemtuzumab, etc；or have treated with thrombopoietin receptor agonist (eg, eltrombopag, romiplostim, rhTPO, etc.) prior to randomization.
3. Previous history of hematopoietic stem cell transplantation.
4. Subjects who is known or suspected of contraindications or hypersensitivity to Hetrombopag's API (Active Pharmaceutical Ingredient).
5. Evidence of clonal cytogenetic abnormalities at the time of screening.
6. Bleeding and/or Infection not adequately responding to appropriate therapy.
7. Any laboratory or clinical evidence for HIV infection. Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subjects screening.
8. ALT> 2.5 x upper limit of normal (ULN), AST> 2.5 x upper limit of normal (ULN) DBLI> 1.5 x upper limit of normal (ULN), Scr> upper limit of normal (ULN).
9. Subjects with uncontrolled hypertension (>180/100mmHg), severe arrhythmia (such as complete left bundle branch block, QT interval prolongation (Bazetts formula), torsade ventricular tachycardia, etc.), unstable angina, pulmonary hypertension at the time of screening.
10. Subjects diagnosed with cirrhosis or portal hypertension.
11. Subjects with malignant solid tumors of any organ system within 5 years prior to screening, with or without treatment, metastasis or recurrence, except for local cutaneous basal cell carcinoma; subjects with hematological tumors found previously or during screening.
12. Subjects with deep vein thrombosis, myocardial infarction, stroke or peripheral arterial embolization within 12 months prior to randomization.
13. Female subjects who are nursing or pregnant.
14. Subjects cannot comply with effective contraception.
15. Subjects have participated in other clinical trial within the 3 months prior to study entry.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Rate of complete hematologic response at six months. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China